CLINICAL TRIAL: NCT01562041
Title: Evaluation of Exercise Treadmill Test Indices in Patients With Cardiovascular Disease
Brief Title: Evaluation of Exercise Treadmill Test (ETT) Indices in Participants With Cardiovascular Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPJMR0032105
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Atherosclerotic Coronary Vascular Disease
Keywords: Cardiovascular disease; Exercise Treadmill Test; Ranolazine; Angina; Myocardial ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Angina Pectoris; Myocardial Ischemia | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ranolazine 500 mg (Experimental): Participants received ranolazine 500 milligrams (mg), orally, twice daily (b.i.d.) up to 14 days.
  Interventions: Drug: Ranolazine 500 mg

INTERVENTIONS:
Drug: Ranolazine 500 mg — Ranolazine 500 mg, oral tablet, b.i.d.
  Other Names: Ranexa®

SUMMARY:
The study was designed to evaluate the use of ETT electrocardiogram (ECG) indices as biomarkers in the assessment of atherosclerotic coronary vascular disease (ASCVD).

ELIGIBILITY:
Inclusion Criteria:

* History of stable coronary artery disease

Exclusion Criteria:

* Inability or unwillingness to participate in multiple exercise treadmill tests and/or any other requirements of this study as assessed by the Investigator.

  * History of chronic atrial fibrillation.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03-09 (Actual); Primary Completion 2014-01-02 (Actual); Study Completion 2014-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 participants took part in the study from 9 March 2012 to 2 January 2014.
Pre-assignment Details: All enrolled participants (N=14) with evidence of exercise induced ischemia [≥ 1 millimeter (mm) ST depression] on the ECG monitoring during exercise treadmill test 1 (ETT 1) and who achieved ≤ 20% variation in exercise duration between consecutive ETTs during baseline period were included in the treatment period. One participant did not provide interpretable treadmill data and was not included in the analysis of primary and secondary variables.
Groups:
- Ranolazine 500 mg: Participants received ranolazine, 500 mg, orally, b.i.d., up to 14 days.
Period: Overall Study
Arm/Group | Ranolazine 500 mg
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants who met the inclusion/exclusion criteria and had at least one post-baseline assessment.
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum ST Segment Change Adjusted for Heart Rate (ST-HR) Index
Description: ST/HR index was measured as the average change in ST segment depression relative to heart rate change over the entire duration of exercise, monitored by ECG during the exercise treadmill tests. Change in maximum ST/HR index between the average of tests 1-3 (pre Ranexa® treatment) performed during baseline period and test 4 (post Ranexa® treatment) during treatment period was reported.
Time Frame: Baseline up to Day 15
Population: Safety Analysis Set included all enrolled participants who met the inclusion/exclusion criteria and had at least one post-baseline assessment. Number analyzed were the number of participants with data available for analysis at given time point.
Measure: Mean (Standard Deviation); unit: microvolts/beats per minute (microV/bpm)
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 13
microvolts/beats per minute (microV/bpm)
  Test 1 | 3.211 (1.6553)
  Test 2 | 2.822 (1.0289)
  Test 3 | 3.228 (1.8910)
  Test 4 | 2.502 (1.8884)
  Change From Baseline in Maximum ST/Heart Rate Index | -0.605 (1.0482)

2. Primary Outcome: Change From Baseline in Maximum ST Segment Change Adjusted for Heart Rate (ST-HR) Slope
Description: ST-HR slope is an index of exercise induced ischemia. Linear regression was used to determine the slope of the ST/HR relationship in a participant's ECG response monitored during the exercise treadmill test. The highest ST segment/heart rate slope from among all the ECG leads and the X-axis intercept of the associated line were used to generate the maximum slope. Change in maximum ST-HR slope between the average of tests 1-3 (pre Ranexa® treatment) performed during baseline period and test 4 (post Ranexa® treatment) during treatment period was reported.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microvolts/beat/minute (microV/beat/min)
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 13
microvolts/beat/minute (microV/beat/min)
  Test 1 | 4.857 (2.3042)
  Test 2 | 5.318 (3.0996)
  Test 3 | 4.645 (2.2869)
  Test 4 | 3.430 (2.7374)
  Change From Baseline in Maximum ST/Heart Rate Slope | -1.553 (3.1200)

3. Primary Outcome: Change From Baseline in X-Axis Intercept of ST-HR Slope
Description: Linear regression was used to determine the slope of the ST/HR relationship in a participant's ECG response monitored during the exercise treadmill test. Change in X- axis intercept of ST-HR slope between the average of tests 1-3 (pre Ranexa® treatment) performed during baseline period and test 4 (post Ranexa® treatment) during treatment period was reported.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 13
beats per minute (bpm)
  Test 1: number analyzed (Participants) | 12
  Test 1 | 93.4 (21.33)
  Test 2 | 88.1 (27.30)
  Test 3 | 89.8 (19.39)
  Test 4: number analyzed (Participants) | 10
  Test 4 | 89.2 (24.34)
  Change From Baseline in X-axis Intercept of ST/Heart Rate Slope: number analyzed (Participants) | 10
  Change From Baseline in X-axis Intercept of ST/Heart Rate Slope | 2.173 (8.7326)

4. Secondary Outcome: Change From Baseline in Total Exercise Duration
Description: Total exercise duration was defined as the elapsed time between the start of exercise and termination of exercise for severe angina, dyspnea or extreme fatigue assessed during the exercise treadmill test. Change in the duration of exercise between the average of tests 1-3 (pre Ranexa® treatment) performed during baseline period and test 4 (post Ranexa® treatment) during treatment period was reported.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 13
minutes
  Test 1 | 11.118 (3.3519)
  Test 2 | 11.008 (3.3765)
  Test 3 | 11.150 (3.4652)
  Test 4 | 11.892 (3.7094)
  Change From Baseline in Total Exercise Duration | 0.755 (0.9834)

5. Secondary Outcome: Change From Baseline in Time to Onset of 1 mm ST Segment Depression (Time to Ischemia)
Description: Exercise-induced ischemia was defined as the new development of horizontal or down sloping ST-segment depression (≥ 1 mm at 60 milliseconds after the J point) vs. baseline tracings. Change in time to onset of 1 mm ST depression between the average of tests 1-3 (pre Ranexa® treatment) performed during baseline period and test 4 (post Ranexa® treatment) during treatment period was reported.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 13
minutes
  Test 1: number analyzed (Participants) | 11
  Test 1 | 8.611 (3.8054)
  Test 2 | 8.833 (3.2241)
  Test 3 | 9.196 (3.6141)
  Test 4: number analyzed (Participants) | 8
  Test 4 | 9.343 (4.1114)
  Change From Baseline in Time to Onset of 1 mm ST Depression: number analyzed (Participants) | 8
  Change From Baseline in Time to Onset of 1 mm ST Depression | 0.876 (1.0227)

6. Secondary Outcome: Change From Baseline in Time to Onset of Angina
Description: Time to onset of angina was defined as the elapsed time between the start of exercise and the onset of anginal chest pain as reported by the participant. Change in time to angina between the average of tests 1-3 (pre Ranexa® treatment) performed during baseline period and test 4 (post Ranexa® treatment) during treatment period was reported.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ranolazine 500 mg
Number analyzed (Participants) | 9
minutes
  Test 1: number analyzed (Participants) | 8
  Test 1 | 8.693 (2.4635)
  Test 2: number analyzed (Participants) | 8
  Test 2 | 7.575 (1.9806)
  Test 3 | 8.189 (1.5457)
  Test 4: number analyzed (Participants) | 7
  Test 4 | 8.037 (3.6395)
  Change From Baseline in Time to Onset of Angina: number analyzed (Participants) | 7
  Change From Baseline in Time to Onset of Angina | 0.473 (3.3342)

ADVERSE EVENTS:
Time Frame: From Baseline up to end of study, approximately 21 days.
Description: Safety analysis set included all participants who received at least one dose of the study drug with at least one post-baseline measurement.
Arm/Group | Ranolazine 500 mg
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine 500 mg (N=14)
NAUSEA (Gastrointestinal disorders) | 1
DIZZINESS (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.